CLINICAL TRIAL: NCT04549129
Title: First Droplets: Feasibility Randomized Controlled Trial of Prenatal Breastfeeding Education
Brief Title: Prenatal Breastfeeding Education
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This pilot study was planned just prior to and during the covid-19 pandemic and was not able to begin due to changes in staffing availability and clinic logistics during the pandemic.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-39614
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Breast Feeding
Keywords: Video education; Hand expression of breast milk; Community health center
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants randomized to the intervention group will receive breastfeeding education and teaching of hand expression using a breastfeeding education video and associated breastfeeding website, as well as hands-on teaching of hand expression techniques during their 36 week visit.
  Interventions: Behavioral: Breastfeeding education video; Behavioral: Breastfeeding website
- Control group (Active Comparator): Participants randomized to the control group will receive usual breastfeeding education during their 36-week visit.
  Interventions: Behavioral: Usual breastfeed education

INTERVENTIONS:
Behavioral: Breastfeeding education video — An introductory video (15 minutes) gives an overview of these "ABCs" (video titled "Term baby" which are further taught through brief text summaries (150-200 words) and short instructional videos (2-6 minutes).
  Arms: Intervention group
Behavioral: Breastfeeding website — The website firstdroplets.com is designed for prenatal education, focusing on the "ABCs of breastfeeding that come before D (delivery)" - attachment (latch), breastmilk production, and calories (transfer of milk to baby).
  Arms: Intervention group
Behavioral: Usual breastfeed education — The usual breastfeed education includes brief counseling by study staff and provision of handouts on latch/positioning and common first week breastfeeding advice
  Arms: Control group

SUMMARY:
In this pilot randomized control trial, the investigators will evaluate the feasibility and acceptability of using a video and website in a prenatal visit to provide breastfeeding education, focusing on how to hand express (HE) breast milk. Participants will be randomized to the video/website intervention group or to the control standard of care group. After delivery, participants will be asked to provide information on how long they breastfed and if they used the information in the video and website. Differences in the outcome measures will be analyzed between the two groups.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility of a new method for teaching breastfeeding skills, and may provide evidence that hand expression (HE) to augment milk production in the first days postpartum can help women breastfeed. Few studies have evaluated the use of HE for improving breastfeeding outcomes. This study will also evaluate the impact of a new video/website which can be utilized widely and adapted for other populations, both in clinical and non-clinical settings.

Prenatal patients receiving care at a community health center in the Boston area will be invited to participate in the study at approximately 28 weeks gestation.

Participants will complete a baseline questionnaire prior to randomization which will occur at the ~36 week prenatal visit. A 1:1 randomization schedule will be applied.

Control arm: participants will be given usual care handouts and the study provider will provide anticipatory guidance and offer to answer any questions about breastfeeding.

Intervention arm: participants will be shown the breastfeeding education video on a study tablet, and provided a QR code which will give them access to the associated website. After watching the video, study staff will then offer to review hand expression by answering questions and reviewing steps, and physically helping the patient to practice hand expression. Hands-on teaching of hand expression will be opt-in only and not required for study participation.

Text messages will be sent to the intervention arm participants with the link to the intervention video and website, and a brief message reminding them to review the materials and to hand express frequently starting immediately after delivery.

All participants (both arms) will be contacted to fill out a very brief, 10-item questionnaire (approximately 5 minutes) at 3 days postpartum, and short questionnaires (10-15 minutes) at 14 days and 60 days postpartum. Questionnaires will ask about use of hand expression, breastfeeding, formula use, perceived breastfeeding problems, breastfeeding efficacy and satisfaction with prenatal breastfeeding education. In all questionnaires participants will be asked about pain and potential adverse events.

Participant and neonatal electronic medical records will reviewed through 2 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Receiving prenatal care at Manet Community Health Center
* Speaks and understands English
* Infants born to the included adult subjects (infants are subjects for chart review only)

Exclusion Criteria:

* Contraindication to breastfeeding (HIV positive or active substance use disorder)
* Fetal demise or neonatal death (after patient is consented into the study)
* Severe maternal illness significant limiting ability to perform hand expression (e.g. admission to ICU during admission for labor and delivery)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Proportion using hand expression | 3 days post partum
  Proportion of respondents who have performed hand expression since their baby was born
Mean times hand expression in past 24 hours | 3 days post partum
  Mean number of times performed hand expression in past 24 hours
Mean hand expression experience scale | 3 days post partum
  Mean score on the following set of questions (adapted from the Breast Milk Expression Experience measure):
  How much do you agree with the following? (1=strongly disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, 5=strongly agree)
  1. My family members support hand expression.
  2. My partner supports hand expression.
  3. I feel peaceful when hand expressing.
  4. I look forward to hand expressing.
  5. I enjoy hand expressing.
  6. Hand expressing is something I could do easily while doing other things.
  7. Hand expressing feels awkward.
  8. Hand expression makes me feel confident my baby is getting enough milk

SECONDARY OUTCOMES:
Proportion exclusively breastfeeding | 2 months
  Proportion who report only giving breastmilk within the past 24 hours
Proportion any breastfeeding | 2 months
  Proportion who report giving any breastmilk within the past 24 hours
Breast feeding self-efficacy | 14 days
  Breast feeding confidence will be assessed using the Breastfeeding Self-Efficacy Scale Short form (BSES-SF) is a 14-item self-administered instrument derived from the original 33-item BSES that measures breastfeeding confidence. All items are preceded by the phrase ''I can always'' and rated on a 5-point Likert scale, ranging from 1 (not at all confident) to 5 (always confident). Scores can range form 14 to 70 and higher scores are associated with higher levels of breast feeding confidence.
Proportion with concern for low milk production | 14 days
  Proportion of mothers who report concern for low milk production
Hand expression comprehension | 36 weeks gestation
  Proportion of correct comprehension of hand expression technique and application after viewing video
Satisfaction with video | 36 weeks gestation
  Mean reported satisfaction with intervention video, on Likert scale (1=Strongly disagree, 2=Disagree, 3=Neither agree nor disagree, 4=Agree, 5=Strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Standish, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Manet Community Health Center, Quincy, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No